CLINICAL TRIAL: NCT05376800
Title: A Phase 0/Ia Study of BI 907828 (Brigimadlin) Concentrations in Brain Tissue and a Non-randomized Open-label, Dose Escalation Study of BI 907828 (Brigimadlin) in Combination With Radiotherapy in Patients With Newly Diagnosed Glioblastoma
Brief Title: A Study to Determine How BI 907828 (Brigimadlin) is Taken up in the Tumor (Phase 0) and to Determine the Highest Dose of BI 907828 (Brigimadlin) That Could be Tolerated (Phase 1a) in Combination With Radiation Therapy in People With a Brain Tumor Called Glioblastoma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 1403-0007; 2023-506409-20-00 (Other: CTIS); 2021-005737-17 (EudraCT Number)
Record Dates: First submitted 2022-05-03; First posted 2022-05-17 (Actual); Last update posted 2025-08-24 (Actual); Status verified 2025-08

CONDITIONS: Glioblastoma
MeSH Terms: conditions — Glioblastoma | interventions — brigimadlin

STUDY DESIGN:
Intervention Model Description: Phase 0 part: measurement of BI 907828 (Brigimadlin) concentrations in brain tissue Phase Ia part: dose escalation
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Phase 0 Part: BI 907828 (Brigimadlin) (Experimental)
  Interventions: Drug: BI 907828 (Brigimadlin)
- Phase Ia Part: BI 907828 (Brigimadlin) (Experimental)
  Interventions: Drug: BI 907828 (Brigimadlin)

INTERVENTIONS:
Drug: BI 907828 (Brigimadlin) — BI 907828 (Brigimadlin)
  Other Names: Brigimadlin

SUMMARY:
This study is open to adults with newly diagnosed glioblastoma, a type of brain tumor. The study has two parts. Part 1 is open to people who can get their brain tumor removed by surgery. Part 2 is open to people who already had such a brain surgery.

This study tests a medicine called BI 907828 (Brigimadlin). BI 907828 (Brigimadlin) is a socalled MDM2 inhibitor that is being developed to treat cancer.

The purpose of Part 1 of the study is to find out how BI 907828 (Brigimadlin) is taken up in the tumor. Participants take a single dose of BI 907828 (Brigimadlin) as a tablet before the brain surgery. Part 1 of the study takes about 1 month. During this time, participants have their brain tumor removed by surgery and visit the study site about 8 times.

The purpose of Part 2 is to find the highest dose of BI 907828 (Brigimadlin) that the participants can tolerate in combination with standard radiation therapy. During the first 6 weeks, participants get standard radiation therapy. In addition, they take a dose of BI 907828 (Brigimadlin) once every 3 weeks. Participants may continue to take BI 907828 (Brigimadlin) as long as they benefit from treatment and can tolerate it. They visit the study site regularly.

During the entire study, doctors also regularly check participants' health and take note of any unwanted effects.

ELIGIBILITY:
Inclusion criteria

* Inclusion criteria Part Phase 0:

  * Histologically (if prior biopsy) or radiologically diagnosed glioblastoma.
  * Neurosurgical tumor resection is indicated and planned according to the assessment of the treating physician.
  * Patients must be at least 18 years old.
  * Eastern Cooperative Oncology Group (ECOG) performance status (PS) of 0 or 1 (an ECOG of 2 is acceptable, if it is due to non-cancer-related disability, and after agreement with the sponsor).
* Inclusion criteria Part Phase Ia:

  * Histologically demonstrated diagnosis of TP53 wild type glioblastoma harboring unmethylated O6-methylguanine-DNA-methyltransferase (MGMT) promoters. Glioblastoma definition according to 2021 World Health Organization (WHO) Classification of Central Nervous System (CNS) tumors, i.e. IDH- wild type only.
  * Patient has undergone neurosurgical tumor resection and is eligible for standard radiotherapy.
  * Patients must be neurologically stable based on the judgement of the treating physician. The use of corticosteroids and anti-seizure medication is allowed and should be at a stable or decreasing dose for at least 7 days before inclusion in the trial. Anti-seizure medication should not include agents that interact with BI 907828 (Brigimadlin).
  * For patients, who have participated in Phase 0, the interval between the single dose of BI 907828 (Brigimadlin) and subsequent Phase 1a treatment must be at least 21 days.

Further inclusion criteria applies.

Exclusion criteria

* Exclusion criteria Part Phase 0:

  * Known TP53 mutant glioblastoma (Note: testing is not mandatory for inclusion).
  * Known Isocitrate dehydrogenase (IDH) mutant grade IV astrocytoma (Note: testing is not mandatory for inclusion).
  * Patient who must receive or intends to receive restricted medications.
  * Patients with pacemakers or other metallic implants that can interfere with the magnetic field during Magnetic Resonance Imaging (MRI) investigations.
  * Inability to undergo contrast-enhanced MRI (Glomerular Filtration Rate (GFR) <30 mL/min).
* Exclusion criteria Part Phase Ia:

  * Patients who have received previous systemic therapy (with the exception of patients who participated in Phase 0) or radiotherapy for glioblastoma.
  * Patients who must or intend to continue the intake of restricted medications or any drug considered likely to interfere with the safe conduct of the trial.
  * Patients with pacemakers or other metallic implants that can interfere with the magnetic field during MRI investigations.
  * Inability to undergo contrast-enhanced MRI (GFR <30 mL/min). Further exclusion criteria applies.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2022-11-30 (Actual); Primary Completion 2025-07-31 (Actual); Study Completion 2025-07-31 (Actual)

PRIMARY OUTCOMES:
Phase 0: Measured total concentration of BI 907828 (Brigimadlin) in brain tissue homogenate from noncontrast enhancing and contrast enhancing brain tumor regions | Up to 24 hours (h)
  Brain tissue samples will be collected after standard of care neurosurgical tumor resection.
  Concentration of BI 907828 (Brigimadlin) will be quantitated in nanomole/kilogram (nmol/Kg) of tissue by validated liquid chromatography mass spectrometry (LC/MS) method.
Phase 0: Calculated unbound concentration of BI 907828 (Brigimadlin) in brain tissue homogenate from noncontrast enhancing and contrast enhancing brain tumor regions | Up to 24 hours (h)
  Brain tissue samples will be collected after standard of care neurosurgical tumor resection.
  Concentration of BI 907828 (Brigimadlin) will be quantitated in nanomole/kilogram (nmol/Kg) of tissue by validated liquid chromatography mass spectrometry (LC/MS) method.
Phase Ia: Occurrence of dose-limiting toxicity (DLT), graded according to Common Terminology Criteria for Adverse Events version 5.0, during the Maximum Tolerated Dose (MTD) evaluation period | Up to 63 Days
Phase Ia: Occurrence of adverse events (AEs) graded according to Common Terminology Criteria for Adverse Events (CTCAE) version 5.0 during the entire treatment period | Up to 7 months.

SECONDARY OUTCOMES:
Phase 0: Dose-dependent changes of expression levels of Tumor suppressor protein p53 (TP53) target genes in contrast enhancing brain regions and non-contrast enhancing brain regions | Up to 24 hours (h)
Phase Ia: Progression-free survival (PFS) | Up to 8 months.
Phase Ia: Maximum plasma concentration (Cmax) of BI 907828 (Brigimadlin) in plasma at Cycle 1 | Up to Day 17
Phase Ia: Area under the Curve of BI 907828 (Brigimadlin) in plasma over the time interval from 0 to the last quantifiable data point (AUC0-tz) | Up to Day 17
Phase Ia: Area under the Curve of BI 907828 (Brigimadlin) in plasma over the time interval from 0 extrapolated to infinity (AUC0-∞) | Up to Day 17

CONTACTS AND LOCATIONS:
Locations (7):
- United States (4):
  - Mayo Clinic-Arizona, Phoenix, Arizona
  - Yale New Haven Hospital, New Haven, Connecticut
  - Mayo Clinic Cancer Center, Jacksonville, Florida
  - Mayo Clinic, Rochester, Rochester, Minnesota
- UZ Leuven, Leuven, Belgium
- Spain (2):
  - Hospital del Mar, Barcelona
  - Hospital Universitario 12 de Octubre, Madrid

IPD SHARING:
Plan to Share IPD: No
Clinical studies sponsored by Boehringer Ingelheim, phases I to IV, interventional and non-interventional, are in scope for sharing of the raw clinical study data and clinical study documents. Exceptions might apply, e.g. studies in products where Boehringer Ingelheim is not the license holder; studies regarding pharmaceutical formulations and associated analytical methods, and studies pertinent to pharmacokinetics using human biomaterials; studies conducted in a single center or targeting rare diseases (in case of low number of patients and therefore limitations with anonymization).
  For more details refer to:
  https://www.mystudywindow.com/msw/datatransparency

REFERENCES:
- See also: Related Info — https://www.mystudywindow.com/